CLINICAL TRIAL: NCT00854126
Title: An Open-label, Phase I, Dose-escalation Study Evaluating GDC-0980 Administered Once Weekly in Patients With Refractory Solid Tumors and Non-hodgkin's Lymphoma
Brief Title: A Study Evaluating GDC-0980 Administered Once Weekly in Patients With Refractory Solid Tumors or Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PIM4605g; MP00881 (Other: Hoffmann-La Roche)
Record Dates: First submitted 2009-02-27; First posted 2009-03-03 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Non-Hodgkin's Lymphoma, Solid Cancers
Keywords: NHL; Solid Tumors; Carcinogenic Tumors
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — 1-(4-((2-(2-aminopyrimidin-5-yl)-7-methyl-4-morpholinothieno(3,2-d)pyrimidin-6-yl)methyl)piperazin-1-yl)-2-hydroxypropan-1-one

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: GDC-0980

INTERVENTIONS:
Drug: GDC-0980 — Escalating repeating dose

SUMMARY:
This is an open-label, multicenter, Phase I study to evaluate the safety, tolerability, and pharmacokinetics of escalating oral doses of GDC-0980 administered to patients with incurable, locally advanced or metastatic solid malignancy or NHL that has progressed or failed to respond to at least one prior regimen or for which there is no standard therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented, incurable, locally advanced or metastatic solid malignancies, or NHL without leukemic phase, that has progressed despite standard of care therapy or for which there is no standard therapy of proven clinical benefit
* A biopsy-accessible lesion from which tissue can be obtained safely
* Evaluable or measurable disease per RECIST and/or the following: prostate cancer patients with non-measurable disease are eligible if they have two rising prostate-specific antigen (PSA) levels that meet the PSA Working Group criteria for progression prior to initiation of study treatment; ovarian cancer patients with non-measurable disease are eligible if they have two rising CA-125 levels greater than the ULN >= 2 weeks apart prior to initiation of study treatment.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 at screening
* Life expectancy >= 12 weeks
* Adequate hematologic and organ function within 28 days before initiation of GDC-0980
* Documented willingness to use an effective means of contraception for both men and women while participating in the study
* For patients participating in DCE-MRI assessments: at least one metastatic lesion measuring >/= 3 cm in the liver or >/= 2 cm elsewhere (lung and mediastinum lesions are ineligible) in at least one dimension (on CT scan)

Exclusion Criteria:

* Leptomeningeal disease as the only manifestation of the current malignancy
* History of Type 1 or 2 diabetes mellitus requiring regular medication
* Grade >=2 hypercholesterolemia or hypertriglyceridemia
* Malabsorption syndrome or other condition that would interfere with enteral absorption
* Known untreated malignancies of the brain or spinal cord, or treated brain metastases that are not radiographically stable for >= 3 months
* Congenital long QT syndrome or screening QTc > 470 msec
* Active congestive heart failure or ventricular arrhythmia requiring medication
* Ejection fraction that is <50% or is below the LLN (whichever is higher), as determined by echocardiogram or MUGA scan
* Active infection requiring IV antibiotics
* Requirement for any daily supplemental oxygen
* DLCO < 50% of predicted value corrected for hemoglobin and alveolar volume
* Uncontrolled hypomagnesemia
* Hypercalcemia requiring continued use of bisphosphonate therapy
* Clinically significant history of liver disease, including viral or other hepatitis, current alcohol abuse, or cirrhosis
* Uncontrolled ascites requiring frequent paracentesis
* Known HIV infection
* Any other diseases, active or controlled pulmonary dysfunction, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or renders the patients at high risk from treatment complications
* Significant traumatic injury within 4 weeks of Day 1
* Major surgical procedure within 4 weeks prior to initiation of GDC-0980
* Treatment with chemotherapy, hormonal therapy (except hormone replacement therapy, oral contraceptives, or GnRH agonists or antagonists for prostate cancer), immunotherapy, biologic therapy, radiation therapy (except palliative radiation to bony metastases), or herbal therapy as cancer therapy within 3 weeks prior to initiation of GDC-0980
* Palliative radiation to bony metastases within 2 weeks prior to initiation of GDC-0980
* Need for chronic corticosteroid therapy of >=10 mg of prednisone per day or an equivalent dose of other anti-inflammatory corticosteroids or immunosuppressant
* Treatment with an investigational agent within 4 weeks prior to initiation of GDC-0980
* Unresolved toxicity from prior therapy except for alopecia and Grade 1 peripheral neuropathy
* Pregnancy or lactation
* For patients participating in DCE-MRI assessments, any contraindication to MRI examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2009-05; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Occurrence of adverse events | Length of study
Occurrence of dose-limiting toxicities | Length of study
Occurrence of Grade 3 and 4 abnormalities in safety-related laboratory parameters and associated dose of GDC-0980 | Length of study
PK parameters after doses of GDC-0980 | Length of study

SECONDARY OUTCOMES:
Best overall response, duration of objective response, and progression-free survival for patients with measurable disease according to RECIST | Length of study
PET response for patients with detectable FDG tumor uptake at baseline | Length of study

CONTACTS AND LOCATIONS:
Overall Officials: Mika Derynck, M.D., Study Director — Genentech, Inc.
Locations (3):
- Boston, Massachusetts, United States
- Villejuif, France
- Manchester, United Kingdom

REFERENCES:
- [Derived] Moein A, Jin JY, Wright MR, Alicke B, Wong H. Retrospective Assessment of Translational Pharmacokinetic-Pharmacodynamic Modeling Performance: A Case Study with Apitolisib, a Dual PI3K/mTOR Inhibitor. Drugs R D. 2024 Jun;24(2):155-167. doi: 10.1007/s40268-024-00459-5. Epub 2024 May 3. PMID 38700808